CLINICAL TRIAL: NCT02357095
Title: Evaluation of the Efficacy and Complications of UACE Combined With Suction Curettage Under Different Kind of Monitoring Methods for the Treatment of Caesarean Scar Pregnancy
Brief Title: UACE Followed by Uterine Suction Curettage for the Treatment of Caesarean Scar Pregnancy
Acronym: UACECSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Yanli Li, Gynecologist, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPT
Record Dates: First submitted 2014-12-29; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Caesarean Scar Pregnancy
Keywords: Caesarean Scar Pregnancy; uterine artery chemo-embolization; treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- hysteroscopic monitoring (Experimental): Method used for the treatment of CSP：Uterine artery chemo-embolization followed by suction curettage under hysteroscopic monitoring.The brand of hysteroscope machine is STORZ.
  Interventions: Procedure: monitoring
- ultrasonography monitoring (Experimental): Method used for the treatment of CSP：Uterine artery chemo-embolization followed by suction curettage under ultrasonography monitoring.The brand of ultrasonograph is mindray(Z6).
  Interventions: Procedure: monitoring
- no monitoring (Experimental): Method used for the treatment of CSP：Uterine artery chemo-embolization followed by suction curettage under no monitoring
  Interventions: Procedure: monitoring

INTERVENTIONS:
Procedure: monitoring — uterine artery chemo-embolization combined with suction curettage under different monitoring methods,such as hysteroscopic monitoring,ultrasonography monitoring and no monitoring

SUMMARY:
The purpose of this study is to determine whether UACE(uterine artery chemo-embolization) followed by suction curettage under the guidance of ultrasonography or hysteroscopy can decrease complications in the treatment of Caesarean scar pregnancy (CSP).

CSP is a special form of ectopic implantation within a fibrous tissue surrounding the previous delivery caesarean scar. The probability of CSP is 1:1800 to 1:2,226 in all pregnancies, and 6.1% in ectopic pregnancy after cesarean delivery. It's a long-term complication after cesarean delivery with very serious consequences,such as uterine rupture and massive uterine bleeding.There are more than ten methods to treat CSP,however, no universal management guidelines have been established up to now.

Present methods for CSP treatment include:1)medical treatment,usually systemic or local methotrexate（MTX）;2）suction curettage;3)medicine combined with uterine curettage;3）surgical treatment（hysteroscopic,laparoscopic or vaginal surgery）;4) uterine artery embolization(UAE);5) The combined use of the above methods.

Moreover, the rupture of the CSP and heavy bleeding may still occur following medical treatment.Suction curettage and excision of the CSP are associated with profuse bleeding. Surgical treatment is less micro-traumatic than nonsurgical interventions. For CSP, UAE followed by suction curettage appears to have more advantage than systemic MTX treatment and may be a priority option.So some author suggests that curettage and systemic methotrexate therapy and embolization as single treatments should be avoided if possible,combination of them is more effective. Plenty of evidences suggested that UACE followed by suction curettage under the guidance of ultrasonography or hysteroscopy is a priority choice.

However,in our clinical practices,suction curettage of CSP is more difficult than usual induced abortion procedure of normal early pregnancy,because PCSD(previous cesarean scar defect)is very common in CSP.In random populations the incidence of PCSD is present in 24%-69% of women evaluated with transvaginal sonography. Scar defects were seen in 61% (66/108), 81% (35/43) and 100% (11/11) of the women who had undergone one, two and at least three Cesarean sections by the transvaginal ultrasound examination.

What is the incidence of complications of suction curettage combined with UACE for CSP treatment remains unknown.How to decrease the complications remains unknown too.So we designed this study.

DETAILED DESCRIPTION:
At first,the investigators evaluated the sample size will be 108 at least through software PASS11, which actually was 144 finally.Then the CSP patients visited or transferred to Maternal and Child Health Hospital of Hubei Province(China) from June 2010 to June 2014 were recruited.Every patient was numbered in chronological sequence.Then participants were randomly assigned into three arms using a randomization table :Group A(Group hysteroscopic monitoring), Group B(Group ultrasonography monitoring),and Group C(Group no monitoring). Randomization was conducted via a system of sealed and numbered envelopes.

Everybody received UACE(uterine artery chemo-embolization) first. Superselective embolization of both uterine arteries was performed using gelatin sponge particles by two experienced radiologists. After the puncture of the right femoral artery, a 5-F Roberts uterine artery catheter was correctly placed in the bilateral uterine artery with the guidance of a 0.889-mm guidewire.A 50mg dose of MTX was infused bilaterally prior to the gelatin sponge particles selective embolism procedure. Postembolization angiography was performed to confirm that the occlusion of the vessels was complete. Within 24-48 h after UACE, women underwent suction curettage.The subatmospheric pressure was 200～500mmHg during suction curettage.

Women assigned to the Group A(Group hysteroscopic monitoring) received UACE followed by suction curettage under hysteroscopic monitoring.Before and after suction curettage, hysteroscopy was performed.If some residual tissues were found, suction curettage would be performed again to remove them.

Women assigned to the Group B(Group ultrasonography monitoring) received UACE followed by suction curettage under ultrasonography monitoring.The suction curettage procedure was performed under abdominal ultrasonography real- time monitoring.When there were nothing residual under ultrasonography,the procedure was completed.

Women assigned to the Group C(Group no monitoring) received UACE followed by suction curettage without monitoring.

All patients were observed during the hospitalization. Ages, weight,gravidity,parity,weeks of gestation, clinical manifestation of CSP,estimated blood loss, operation time,length of uterine cavity and PCSD(previous cesarean scar defect), and side effects(such as fever, nausea,and low abdominal pain) were recorded. The serum β-hCG level and renal, hepatic function, and complete blood count were measured before intervention. The size of the gestation sac or a heterogeneous mass was measured by transvaginal ultrasound at the same time.

The patients were followed up by measuring serum β-hCG level every week until the β-hCG level reverted to normal.All women were followed up 2 weeks and 2 months after operation, which included ultrasound examination, and clinical assessment (bleeding pattern and resumption of menses).

Theχ2 test were used for the analysis of enumeration data. The measurement data comparisons between groups were tested by ANOVA analysis. A probability value of<.05 was considered statistically significant.All data analyses were conducted with SPSS software (version17.0;SPSS,Inc,IBM,American).

ELIGIBILITY:
Inclusion Criteria:

* pre-operative diagnosed as CSP;hemodynamic stability

Exclusion Criteria:

* acute PID(pelvic inflammatory disease) or vaginitis;shock;prior classical cesarean section;prior treatment with suction curettage or MTX

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The number of participants with complications in different Arms. | two months
  The complications of blood loss,incomplete abortion,intrauterine adhesions,induced abortion syndrome,uterine perforation,PID,and amnionic fluid embolism are recorded.The number of participants with complications in different Arms is counted.
Composite outcome measure：the effectiveness of UACE followed by suction curettage for the treatment of CSP | two months
  Serum hCG are measured every week post-operation till it resolute to normal level.Operation time are recorded.The time of menstrual recovery are recorded.

SECONDARY OUTCOMES:
Composite outcome measure：Baseline clinical characteristic of patient when diagnosed with CSP | one week
  Age,body weight,gravity and parity,previous caesarean section times,interval from last caesarean section,gestation age and symptoms when diagnosed,pre-treatment human chorionic gonadotropin(hCG) level and size of gestational sac are collected to investigate the relation between these index and CSP

CONTACTS AND LOCATIONS:
Overall Officials: Wu X-Feng, Ph.D & MD, Study Chair — Maternal and Child Health Hospital of Hubei Province,Wuhan,Hubei,PR China; Gao Han, Bachelor, Principal Investigator — Maternal and Child Health Hospital of Hubei Province,Wuhan,Hubei,PR China; Ma Quan-Fu, Ph.D & MD, Study Director — Maternal and Child Health Hospital of Hubei Province,Wuhan,Hubei,PR China

REFERENCES:
- [Result] Jurkovic D, Hillaby K, Woelfer B, Lawrence A, Salim R, Elson CJ. First-trimester diagnosis and management of pregnancies implanted into the lower uterine segment Cesarean section scar. Ultrasound Obstet Gynecol. 2003 Mar;21(3):220-7. doi: 10.1002/uog.56. PMID 12666214
- [Result] Stevens EE, Ogburn P. Cesarean scar ectopic pregnancy: a case report of failed combination local and systemic methotrexate management requiring surgical intervention. J Reprod Med. 2011 Jul-Aug;56(7-8):356-8. PMID 21838169
- [Result] Wang CJ, Yuen LT, Chao AS, Lee CL, Yen CF, Soong YK. Caesarean scar pregnancy successfully treated by operative hysteroscopy and suction curettage. BJOG. 2005 Jun;112(6):839-40. doi: 10.1111/j.1471-0528.2005.00532.x. No abstract available. PMID 15924549
- [Result] Zhuang Y, Huang L. Uterine artery embolization compared with methotrexate for the management of pregnancy implanted within a cesarean scar. Am J Obstet Gynecol. 2009 Aug;201(2):152.e1-3. doi: 10.1016/j.ajog.2009.04.038. Epub 2009 Jun 13. PMID 19527897
- [Result] Timor-Tritsch IE, Monteagudo A. Unforeseen consequences of the increasing rate of cesarean deliveries: early placenta accreta and cesarean scar pregnancy. A review. Am J Obstet Gynecol. 2012 Jul;207(1):14-29. doi: 10.1016/j.ajog.2012.03.007. Epub 2012 Mar 10. PMID 22516620
- [Result] Zhuang YL, Wei LH, Wang W, Huang LL. [Treatment of pregnancy in a previous caesarean section scar with uterine artery embolization: analysis of 60 cases]. Zhonghua Yi Xue Za Zhi. 2008 Aug 26;88(33):2372-4. Chinese. PMID 19087704
- [Result] Lan W, Hu D, Li Z, Wang L, Yang W, Hu S. Bilateral uterine artery chemoembolization combined with dilation and curettage for treatment of cesarean scar pregnancy: A method for preserving the uterus. J Obstet Gynaecol Res. 2013 Jun;39(6):1153-8. doi: 10.1111/jog.12051. Epub 2013 May 30. PMID 23718134
- [Result] Zhang XB, Zhong YC, Chi JC, Shen JL, Qiu XX, Xu JR, Zhao AM, Di W. Caesarean scar pregnancy: treatment with bilateral uterine artery chemoembolization combined with dilation and curettage. J Int Med Res. 2012;40(5):1919-30. doi: 10.1177/030006051204000533. PMID 23206476
- [Result] van der Voet LF, Vervoort AJ, Veersema S, BijdeVaate AJ, Brolmann HA, Huirne JA. Minimally invasive therapy for gynaecological symptoms related to a niche in the caesarean scar: a systematic review. BJOG. 2014 Jan;121(2):145-56. doi: 10.1111/1471-0528.12537. PMID 24373589
- [Result] Osser OV, Jokubkiene L, Valentin L. High prevalence of defects in Cesarean section scars at transvaginal ultrasound examination. Ultrasound Obstet Gynecol. 2009 Jul;34(1):90-7. doi: 10.1002/uog.6395. PMID 19499514
- [Derived] Li Y, Gong L, Wu X, Gao H, Zheng H, Lan W. Randomized controlled trial of hysteroscopy or ultrasonography versus no guidance during D&C after uterine artery chemoembolization for cesarean scar pregnancy. Int J Gynaecol Obstet. 2016 Nov;135(2):158-162. doi: 10.1016/j.ijgo.2016.04.019. Epub 2016 Aug 5. PMID 27634054